CLINICAL TRIAL: NCT01702493
Title: A Phase 1, Open-Label, Randomized, Controlled, Four-Period Crossover Study to Assess the Relative Bioavailability of New Oral Formulations of SRT2104 in Healthy Male Volunteers
Brief Title: A Study to Assess the Relative Bioavailability of New Oral Formulations of SRT2104 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 117041
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Psoriasis
Keywords: SRT2104; Modified Release; Bioavailability; Crossover
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1: Cap SRT2104 (Active Comparator): 500 mg SRT2104 (in the form of two, 250 mg capsules) will be administered as a single oral dose in the fasting state
  Interventions: Drug: Cap SRT2104
- Part 1: Tab SRT2104 (slow release) (Experimental): 500 mg SRT2104 (in the form of two, 250 mg slow release tablets) will be administered as a single oral dose in the fasting state.
  Interventions: Drug: Tab SRT2104 slow release
- Part 1: Tab SRT2104 (intermediate release) (Experimental): 500 mg SRT2104 (in the form of two, 250 mg intermediate release tablets) will be administered as a single oral dose in the fasting state.
  Interventions: Drug: Tab SRT2104 intermediate release
- Part 1: Tab SRT2104 (fast release) (Experimental): 500 mg SRT2104 (in the form of two, 250 mg fast release tablets) will be administered as a single oral dose in the fasting state.
  Interventions: Drug: Tab SRT2104 fast release
- Part 2A: SRT2104 500 mg single-dose (Experimental): 500 mg SRT2104 (formulation selected from Part 1) will be administered as a single oral dose in the fed state.
  Interventions: Drug: Selected formulations of SRT2104 from Part 1
- Part 2B: SRT2104 single alternative dose (Experimental): An alternative dose (other than 500 mg, but not to exceed 2000 mg) of SRT2104 (formulation selected from Part 1) will be administered as a single oral dose.
  Interventions: Drug: Selected formulations of SRT2104 from Part 1 single alternative dose
- Part 2C: SRT2104 500 mg daily for 7 days (Experimental): 500 mg SRT2104 (formulation selected from Part 1) will be administered daily for 7 days.
  Interventions: Drug: Selected formulations of SRT2104 from Part 1

INTERVENTIONS:
Drug: Cap SRT2104 — Micronized free base in a 250 mg SRT2104 (active equivalents) capsule
  Arms: Part 1: Cap SRT2104
Drug: Tab SRT2104 slow release — New 250 mg SRT2104 mesylate salt slow release tablet
  Arms: Part 1: Tab SRT2104 (slow release)
Drug: Tab SRT2104 intermediate release — New 250 mg SRT2104 mesylate salt intermediate release tablet
  Arms: Part 1: Tab SRT2104 (intermediate release)
Drug: Tab SRT2104 fast release — New 250 mg SRT2104 mesylate salt fast release tablet
  Arms: Part 1: Tab SRT2104 (fast release)
Drug: Selected formulations of SRT2104 from Part 1 — SRT2104 500 mg of selected formulation(s) from Part 1 in single-dose or daily for 7 days
  Arms: Part 2A: SRT2104 500 mg single-dose; Part 2C: SRT2104 500 mg daily for 7 days
Drug: Selected formulations of SRT2104 from Part 1 single alternative dose — SRT2104 single alternative dose (other than 500 mg, but not to exceed 2000 mg) of selected formulation(s) from Part 1
  Arms: Part 2B: SRT2104 single alternative dose

SUMMARY:
This is an open-label, randomized, controlled, single center study to assess the safety, variability in exposure, and relative bioavailability of new oral formulations of SRT2104. This is a two part study and each part consists of screening (within 21 days of the first scheduled dose of SRT2104), treatment period and follow-up visit (approximately 6 days after the last dose). Part 1: Subjects will receive all four fomulations of SRT2104 and their order of their doses will be randomized. Each subject will receive one formulation as a 500 milligram (mg) dose (in the form of two 250 mg capsules or tablets) in each session given in the fasted state. Each dose will be separated by at least 6 days. Pharmacokinetic (PK) sampling will be done pre and post each scheduled dosing session. After all 4 dosing sessions, the safety and PK data will be reviewed to determine which, if any, formulation(s) will be carried forward into Part 2. The total duration will be approximately 7 weeks. Part 2: Is further divided into Part 2A, 2B and 2C of the study and are optional. After the completion of Part 1, the sponsor will decide whether to proceed with any or all of Part 2, and whether the selected formulation(s) is to be administered in the fed or fasted state for Parts 2B and 2C. For all the sub parts of Part 2 the pre and post-dose PK samples will be obtained. Part 2A: A single-dose of the selected formulation(s) from Part 1 will be administered after a standard meal to assess the effect of food on the bioavailability of SRT2104 at the 500 mg dose. The total duration will be approximately 4 weeks. Part 2B: A single alternative dose (other than 500 mg, but not to exceed 2000 mg) of the selected formulation(s) from Part 1 will be administered to assess the safety and PK profile of this dose level. The total duration will be approximately 4 weeks. Part 2C: The selected formulation(s) from Part 1 will be administered at the 500 mg dose once daily for 7 consecutive days, to assess the safety and tolerability and characterize the PK profile of repeat dosing. The total duration will be approximately 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician.
* Males between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight >=50 kilogram (kg) (110 lbs) and body mass index (BMI) >=18.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Past or present disease that is judged by the investigator to have the potential to interfere with the study procedures or compromise the subject's safety.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), or aspartate aminotranferase (AST), alanine aminotranferase (ALT), alkaline phosphatase and bilirubin >1.5 x upper limit of normal (ULN).
* Abnormalities on the Screening or Day -1: electrocardiogram (ECG) that, in the opinion of the investigator, will compromise subject safety in the study or QT corrected using Fridericia's formula (QTcF) > 450 milliseconds (msec).
* A history of Hepatitis B, Hepatitis C or human immunodeficiency virus (HIV), or positive serology at Screening.
* History of regular alcohol consumption within 6 months of the Screening (Screening visit) and a positive pre-study drug/alcohol screen.
* Participation in a clinical trial and treatment with an investigational product within 3 months prior to Screening visit.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Where participation in the study would result in the inability to donate blood or blood products in excess of 500 milliliter (mL) within a 56 day period.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10-30 (Actual); Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-05 (Actual)

PRIMARY OUTCOMES:
Measure of variability in exposure-CVw | Part 1: Days 1, 8, 15 and 22; Parts 2A and 2B: Day 1; Part 2C: Days 1 to 7. Pre dose and post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after each scheduled dosing session.
  The variability in exposure of SRT2104 will be assessed by calculating the within subject coefficient of variation (CVw).
Measure of relative bioavailability-AUC | Part 1: Days 1, 8, 15 and 22; Parts 2A and 2B: Day 1; Part 2C: Days 1 to 7. Pre dose and post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after each scheduled dosing session.
  Relative bioavailability of SRT2104 will be assessed by evaluating area under the curve (AUC).
Measure of relative bioavailability-Cmax | Part 1: Days 1, 8, 15 and 22; Parts 2A and 2B: Day 1; Part 2C: Days 1 to 7. Pre dose and post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after each scheduled dosing session.
  Relative bioavailability of SRT2104 will be assessed by measuring maximum observed plasma concentration (Cmax).
Measure of relative bioavailability-Tmax | Part 1: Days 1, 8, 15 and 22; Parts 2A and 2B: Day 1; Part 2C: Days 1 to 7. Pre dose and post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after each scheduled dosing session.
  Relative bioavailability of SRT2104 will be assessed by measuring the time to reach maximum observed plasma concentration (Tmax).
Safety of SRT2104 as assessed by number of subjects with adverse events (AE)s | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety parameter will include recording number of AEs, throughout the study.
Safety of SRT2104 as assessed by intensity of AEs | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety parameter will include recording of intensity of AEs, throughout the study.
Safety of SRT2104 as assessed by type of AEs | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety parameter will include recording of type of AEs, throughout the study.
Safety of SRT2104 as assessed by change from Baseline in heart rate | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety will be assessed by recording heart rate at Baseline and at end of the study.
Safety of SRT2104 as assessed by change from Baseline in blood pressure | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety will be assessed by recording blood pressure at Baseline and at end of the study.
Safety of SRT2104 as assessed by change from Baseline in temperature | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety will be assessed by recording temperature at Baseline and at end of the study.
Safety of SRT2104 as assessed by change from Baseline in ECG readings | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Safety will be assessed by recording the electrocardiogram (ECG) readings at Baseline and at end of the study.
Safety of SRT2104 as assessed by change from Baseline in clinical laboratory parameters | Part 1: 7 weeks; Part 2A: 4 weeks; Part 2B: 4 weeks; Part 2C: 5 weeks.
  Clinical laboratory parameters will include hematology, clinical chemistry and electrolytes, serology, coagulation and urinalysis. Safety will be assessed by evaluating the clinical laboratory parameter readings at Baseline and at end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 117041 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117041?search=study&study_ids=117041#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117041 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register